CLINICAL TRIAL: NCT03340480
Title: The Food Effect on the Pharmacokinetics of NVP-1402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: NVP-1402-02
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1402-1 (Experimental): NVP-1402 was administered once a day for 24 hours
  Interventions: Drug: NVP-1402
- NVP-1402-2 (Experimental): NVP-1402 was administered once a day for 24 hours
  Interventions: Drug: NVP-1402

INTERVENTIONS:
Drug: NVP-1402 — Oral

SUMMARY:
The purpose of this study is to evaluate the food effect on the pharmacokinetics of NVP-1402 in healthy male volunteers.

DETAILED DESCRIPTION:
This study is designed as randomized, open-label, single oral dose, two-treatment, two sequence crossover active-controlled and crossover assignment for evaluate the food effect on the pharmacokinetics of NVP-1402 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* No history of clinically significant medical disorder
* Capable of consent to participate in the study

Exclusion Criteria:

* History of hypersensitive reactions to study drug or other related drugs
* Any significant abnormality found during screening
* Any significant medical history
* History of alcohol abuse, smoking continuously
* History of drug abuse
* Clinically significant surgery within 4 weeks prior to administration of the study drug
* Participation in another clinical trial within 3 months prior to administration of the study drug

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma: Cmax | up to 24 hours after administration
  Maximum measured concentration of the analyte in plasma
Pharmacokinetics of plasma: AUClast | up to 24 hours after administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point

SECONDARY OUTCOMES:
Pharmacokinetics of plasma: AUCinf | up to 24 hours after administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity
Pharmacokinetics of plasma: Tmax | up to 24 hours after administration
  Time from dosing to the maximum measured concentration of the analyte in plasma
Pharmacokinetics of plasma: t1/2 | up to 24 hours after administration
  Terminal half-life of the analyte in plasma

CONTACTS AND LOCATIONS:
Overall Officials: D Seong Shin, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Navipharm, Suwon, Gyeonggi-do, South Korea